CLINICAL TRIAL: NCT00437034
Title: A Phase 2 Study of Aflibercept for the Treatment of Relapsed or Refractory Multiple Myeloma
Brief Title: Aflibercept for Relapsed Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00181; NCI-2009-00181 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0608008688 (Other: Montefiore Medical Center); 7521 (Other: CTEP/NCI); P30CA013330 (NIH); N01CM62204 (NIH)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Results first posted 2015-07-29 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (antiangiogenesis therapy) (Experimental): Patients receive aflibercept IV over 1 hour on day 1. Treatment repeats every 2 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: aflibercept

INTERVENTIONS:
Biological: aflibercept — Given IV
  Other Names: vascular endothelial growth factor trap; VEGF Trap; Zaltrap

SUMMARY:
This phase II trial is studying the side effects and how well aflibercept works in treating patients with stage II or stage III multiple myeloma that has relapsed or not responded to previous treatment. Aflibercept may be able to carry cancer-killing substances directly to multiple myeloma cells. It may also stop the growth of multiple myeloma by blocking blood flow to the cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To evaluate the safety and efficacy of VEGF Trap (aflibercept) in patients with relapsed or refractory, stage II or III multiple myeloma (MM).

II. To perform correlative studies in order to evaluate the angiogenic properties of tissue from patients during the course of treatment with VEGF Trap.

OUTLINE: This is a multicenter study.

Patients receive aflibercept intravenously (IV) over 1 hour on day 1. Treatment repeats every 2 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 60 days and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed multiple myeloma

  * Stage II or III disease according to Salmon-Durie staging criteria
* Relapsed or refractory disease
* Progressive disease
* Measurable disease, defined by ≥ 1 of the following criteria:

  * Serum M protein ≥ 1.0 g/dL by serum protein electrophoresis
  * Free light chain measurement > 200 mg/dL
  * Urinary M protein excretion ≥ 200 mg/24 hours
* Must have received ≥ 2 prior therapies* for multiple myeloma that meet the following criteria:

  * Antimyeloma therapeutic regimen consisting of ≥ 1 complete course of single-agent or combination-agent therapy, or a planned series of treatments (e.g., 3-4 courses of induction therapy followed by a stem cell harvest procedure followed by conditioning high-dose therapy supported by stem cell transplantation)
  * Antimyeloma regimen is discontinued because of the development of resistant disease or severe therapy-related toxicity
  * Individual antimyeloma regimen will be considered to have been discontinued when all agents of the regimen have been permanently stopped
  * A prior regimen will not be considered to have been discontinued for the modification of drug doses, or if less than all the agents of a combination regimen have been discontinued, or if the regimen has been halted temporarily for the development of a plateau phase of myeloma
  * Maintenance therapy will not be considered an additional regimen
  * If new agents are added to an existing regimen, presumably because of tumor resistance, the old regimen will be considered to have ended and a new regimen to have started
* No evidence of central nervous system (CNS) disease, including primary brain tumor or brain metastasis
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 12 weeks
* White blood cell (WBC) ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 75,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times ULN
* Creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 60 mL/min
* No albuminuria only

  * Urine protein: creatinine ratio < 1 OR 24-hour urine protein with an albumin level < 500 mg
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study therapy

Exclusion criteria:

* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No known history of allergic reactions attributed to compounds of similar chemical or biological composition to other agents used in the study
* No serious or nonhealing wound, ulcer, or bone fracture
* No significant traumatic injury within the past 28 days
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No clinically significant cardiovascular disease
* No prothrombin time (PT) or international normalized ratio (INR) > 1.5 (unless patient is on full-dose warfarin)
* No evidence of bleeding diathesis or coagulopathy
* No uncontrolled intercurrent illness that would limit compliance with study requirements, including ongoing or active infection
* No psychiatric illness or social situations that would limit study compliance
* No concurrent major surgery
* No concurrent immunosuppressive agents (including steroids)
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-01; Primary Completion 2010-10 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Niesvizky-Iszaevich, Principal Investigator — Montefiore Medical Center
Locations (6):
- United States (6):
  - North Shore University Hospital, Manhasset, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 6 patients were enrolled at two institutions between January 2007 and April 2010
Period: Overall Study
Arm/Group | Treatment (Antiangiogenesis Therapy)
Started | 6
Completed | 0
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Disease progression during treatment | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Antiangiogenesis Therapy)
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 59 [37 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race/Ethnicity, Customized [Number; unit: participants]
  White | 4
  African American | 1
  Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete [CR] and Partial Response [PR])
Description: A 95% confidence interval was intended to be estimated via binomial proportions, but was not computed due to small sample size.
  Criteria for Response from EBMT, IBMTR, ABMTR: Complete Response:Complete absence of monoclonal protein by immunofixation for a minimum of 6 weeks; Near Complete Response:Absence of serum paraprotein by standard serum/urine protein electrophoresis without disappearance of monoclonal spike by immunofixation; Partial Response:Sustained decrease in production rate of monoclonal serum protein to 50% or less of pretreatment value; Stable Disease: No significant change from baseline; Progression of Disease:Patients with a > or = 25% rise in production rate, new/increased size of lytic lesions/plasmacytomas/progressive marrow plasmacytosis; Symptomatic Deterioration:Patients with deterioration of health requiring discontinuation of treatment w/out objective evidence of disease progression.
Time Frame: At baseline and every 4 weeks during study treatment until treatment discontinuation due to disease progression, unacceptable toxicities and/or patient withdrawal.
Measure: Number; unit: participants
Arm/Group | Treatment (Antiangiogenesis Therapy)
Number analyzed (Participants) | 6
participants
  Disease progression | 5
  Stable disease | 1

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Assessed by Kaplan-Meier survival analysis and 95% confidence intervals will be calculated using Greenwood's formulae.
Time Frame: Time from first treatment day until objective or symptomatic progression, assessed up to 6 months
Population: Data not collected
Arm/Group | Treatment (Antiangiogenesis Therapy)
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival (OS)
Description: Assessed by Kaplan-Meier survival analysis and 95% confidence intervals will be calculated using Greenwood's formulae.
Time Frame: Time from first treatment day until death, assessed up to 6 months
Population: Overall survival was not assessed by the Kaplan-Meier survival or calculated using the Greenwood's formulae.
Arm/Group | Treatment (Antiangiogenesis Therapy)
Number analyzed (Participants) | 0

4. Secondary Outcome: Toxicities
Description: Toxicities will be assessed and graded according to Common Terminology Criteria for Adverse Events (CTCAE) v. 3.0 terminology. Exact 95% confidence intervals around the toxicity proportions will be calculated to assess the precision of the obtained estimates.
Time Frame: up to 6 months
Population: Participants with grade 1 and 2 adverse events
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Antiangiogenesis Therapy)
Number analyzed (Participants) | 6
Participants | 6

5. Secondary Outcome: Tissue Expression Patterns of VEGFR Subtypes
Description: The change in the prevalence/expression of these markers between pre-and-post treatment samples will be analyzed by McNemar's test. Ninety-five percent confidence intervals will be calculated to assess the precision of the obtained estimates for all laboratory correlates.
Time Frame: At baseline and post-treatment (1 week after 2nd dose and end of study)
Population: data not collected
Arm/Group | Treatment (Antiangiogenesis Therapy)
Number analyzed (Participants) | 0

6. Secondary Outcome: The Apoptotic State of Tumor Neovasculature
Description: as for outcome 5
Time Frame: At baseline and post-treatment (1 week after 2nd dose and end of study)
Population: data not collected
Arm/Group | Treatment (Antiangiogenesis Therapy)
Number analyzed (Participants) | 0

7. Secondary Outcome: Proangiogenic Factors Such as VEGF
Description: as for outcome 5
Time Frame: At baseline, before every course for 3 months, and then every 3 months during treatment for the first year
Population: data not collected
Arm/Group | Treatment (Antiangiogenesis Therapy)
Number analyzed (Participants) | 0

8. Secondary Outcome: Circulating Endothelial Progenitors
Description: as for outcome 5
Time Frame: At baseline, before every course for 3 months, and then every 3 months during treatment for the first year
Population: data not collected
Arm/Group | Treatment (Antiangiogenesis Therapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Antiangiogenesis Therapy)
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Antiangiogenesis Therapy) (N=6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypertension (Vascular disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1)
ODYNOPHAGIA (PAINFUL SWALLOWING) (Gastrointestinal disorders) | 1 (1)
Voice changes (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash: desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Pain: Muscle (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Leukocytes decreased (Investigations) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less